CLINICAL TRIAL: NCT06317675
Title: Osteopathic Manipulative Treatment for Patients Affected by Symptoms Related to Gastro-oesophageal Reflux Disease
Brief Title: Osteopathic Manipulative Treatment for Gastro-oesophageal Reflux Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Studio Osteopatico Busto Arsizio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ct9873
Record Dates: First submitted 2024-02-29; First posted 2024-03-19 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Gastro-oesophageal Reflux Disease
Keywords: GERD; Osteopathic manipulative treatment; OMT; Manual therapy
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Manipulation, Osteopathic; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Osteopathic manipulative treatment (OMT) (Experimental): Participants will receive four OMTs at week 1, 2, 4 and 8. Joint mobilization techniques for ribs, cervical and dorsal spine, as well as visceral treatment, soft-tissue release on diaphragm and abdominal wall will be used.
  Interventions: Other: Osteopathic manipulative treatment (OMT)
- OMT + breathing exercises. (Active Comparator): This group will receive OMTs and five breathing exercises to perform daily at home. A recorded video of the exercises will be provided to participants in this group.
  Interventions: Other: Osteopathic manipulative treatment (OMT)
- Control (No Intervention): Usual care group (PPI or reflux suppressant)

INTERVENTIONS:
Other: Osteopathic manipulative treatment (OMT) — Manual therapy on different area of the body.
  Other Names: Manipulative treatment; Manual therapy
  Arms: OMT + breathing exercises.; Osteopathic manipulative treatment (OMT)

SUMMARY:
To evaluate the effects of osteopathic manipulative treatment in patients affected by symptoms related to gastro-oesophageal reflux disease (GERD)

ELIGIBILITY:
Inclusion Criteria:

* Retrosternal burning sensation and/or regurgitation
* Diagnosis of reflux with any methodology
* Duration of symptoms for more than 3 months
* Taking short or long-term proton pump inhibitors (as needed, treatment start date and expected end date, mg, drug name)
* With or without esophagitis
* With or without hiatal hernia
* With or without helicobacter pylori
* GERDQ questionnaire > 8 points

Exclusion Criteria:

* neoplastic pathologies
* patients who have undergone surgery for GERD
* systemic pathologies (rheumatic, infectious conditions, feverish state, vascular alterations, endocrine diseases including diabetes, metabolic and neoplastic syndromes),
* patients already undergoing manipulative therapy for reflux
* patients with active gastric ulcers
* congenital or acquired immune diseases
* allergic state of any kind
* pregnancy
* use of intrauterine device
* patients undergoing corticosteroid therapy
* patients already subjected to manual/respiratory therapy in the last 3 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Mean change in GERD-HRQL | At week 2, 4 an 8.
  best possible score: 0, worst possible score: 50
Adverse effects | At week 2, 4 and through study completion (8 weeks)
  Type and number.

SECONDARY OUTCOMES:
Exercise adherence | through study completion (8 weeks)
  number of exercises per day performed by participants in OMT + exercise group.
Change in drugs use | At week 2, 4 and 8.
  Types, number and frequency of drug assumptions (such as PPI and other oral suspensions)

CONTACTS AND LOCATIONS:
Locations (1):
- CTFO, Saronno, Varese, Italy

IPD SHARING:
Plan to Share IPD: No